CLINICAL TRIAL: NCT00225745
Title: Assessment of Plasma Ghrelin Levels in Patients With Pancreatic Cancer
Brief Title: Ghrelin Levels in Pancreatic Cancer Patients
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: DMS 0405
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-08

CONDITIONS: Pancreatic Cancer
Keywords: Ghrelin
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Whole Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Pancreatic cancer patients
  Interventions: Procedure: Blood draw
- 2: Healthy controls
  Interventions: Procedure: Blood draw

INTERVENTIONS:
Procedure: Blood draw — One blood draw prior to first treatment

SUMMARY:
The primary outcome measure for this study is plasma ghrelin level.

DETAILED DESCRIPTION:
The primary outcome measure for this study is plasma ghrelin level, and the two primary comparison are:

* Patients with cachexia versus patients without cachexia
* Patients with cachexia versus healthy controls

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of pancreatic adenocarcinoma
* The control are will include healthy age-matched patients without cancer
* The test arm will include patients with pancreatic cancer and they will divided into two groups: those with and without weight loss
* Patients must have recovered from any major infections and/or surgical procedures

Exclusion Criteria:

* Patients with other serious medical illness like congestive heart failure, thyroid disease,liver disease or renal failure - conditions that will alter their nutritional state
* Patients on appetite stimulant and those receiving total parenteral nutrition
* Patients who have undergone gastrectomy or those who have gastric ulcers
* Patients receiving active chemotherapy
* No prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer or for which patient has been disease free for at least five years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pancreatic cancer patients who have not received treatment. Healthy age-matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2004-04; Primary Completion 2013-10 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
To evaluate plasma ghrelin levels in patients with pancreatic cancer and compare with age matched controls | prior to treatment

SECONDARY OUTCOMES:
To investigate the role of ghrelin in pathophysiology of cancer cachexia | prior to treatment
To generate hypotheses for future studies and treatment based on the findings | prior to treatment

CONTACTS AND LOCATIONS:
Overall Officials: J Marc Pipas, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center/Norris Cotton Cancer Center, Lebanon, New Hampshire, United States